CLINICAL TRIAL: NCT05643066
Title: Discharge Readiness After Propofol With or Without Esketamine for Outpatient Flexible Bronchoscopy: a Randomized, Controlled Study
Brief Title: Esketamine-propofol Versus Propofol for Flexible Bronchoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Yao Yusheng, Clinical Professor, Fujian Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K2021-12-067
Record Dates: First submitted 2022-11-14; First posted 2022-12-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Recovery
Keywords: bronchoscopy; esketamine; procedure sedation; propofol
MeSH Terms: interventions — Esketamine; Saline Solution; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.1 mg/kg esketamine group (Experimental): Procedure sedation was induced using intravenous 0.1 mg/kg esketamine and propofol 1 mg/kg. Afterward, propofol 0.5 mg/kg was administered to maintain the target sedation level (MOAA/S of less than three).
  Interventions: Drug: 0.1 mg/kg esketamine; Drug: Propofol
- 0.2 mg/kg esketamine group (Experimental): Procedure sedation was induced using intravenous 0.2 mg/kg esketamine and propofol 1 mg/kg. Afterward, propofol 0.5 mg/kg was administered to maintain the target sedation level (MOAA/S of less than three).
  Interventions: Drug: 0.2 mg/kg esketamine; Drug: Propofol
- Placebo group (Placebo Comparator): Procedure sedation was induced using intravenous 0.9% saline and propofol 1 mg/kg. Afterward, propofol 0.5 mg/kg was administered to maintain the target sedation level (MOAA/S of less than three).
  Interventions: Drug: 0.9% saline; Drug: Propofol

INTERVENTIONS:
Drug: 0.1 mg/kg esketamine — Esketamine 0.1 mg/kg was intravenously injected first.
  Other Names: S-ketamine 0.1 mg/kg
  Arms: 0.1 mg/kg esketamine group
Drug: 0.2 mg/kg esketamine — Esketamine 0.2 mg/kg was intravenously injected first.
  Other Names: S-ketamine 0.2 mg/kg
  Arms: 0.2 mg/kg esketamine group
Drug: 0.9% saline — 0.9% saline was intravenously injected first.
  Other Names: Normal saline
  Arms: Placebo group
Drug: Propofol — Propofol 1 mg/kg was injected immediately. Afterward, propofol 0.5 mg/kg was administered to maintain the target sedation level (MOAA/S of less than three).
  Other Names: propofol injection

SUMMARY:
Bronchoscopy is a promising technology for lung and bronchus disease detection and therapy. However, this procedure is associated with a relatively high risk of hypoxemia, coughing, wheezing, and dyspnea. Despite the fact that propofol is the most commonly used agent in procedure sedation, the narrow therapeutic index remains challenging. Esketamine is the s-enantiomer of ketamine with potent analgesic and sedative properties. This study aims to test the hypothesis that adding subanesthetic esketamine to propofol is non-inferior to propofol alone for bronchoscopy on the recovery profile and discharge from the hospital.

DETAILED DESCRIPTION:
Bronchoscopy is one of the most common procedures to detect lung and bronchus disease. The procedure is generally uncomfortable and associated with a relatively high risk of hypoxemia, coughing, wheezing, and dyspnea. Therefore, physicians are placing increasing importance on the use of procedure sedation due to the demand for comfortable medical care.

Propofol is an effective agent for sedation in bronchoscopy with rapid onset and recovery. However, the safety endpoints of propofol are not cost-effective, including injection pain, hypotension, apnea, airway compromise, and without a reversal agent. Specifically, the depressive effects on the respiratory system are more noteworthy in bronchoscopy, which may lead to hypoxia. These drawbacks may hinder functional recovery and delay the discharge time. Hence, physicians are searching for an optimal sedation regimen for bronchoscopy.

Esketamine, the s-enantiomer of ketamine, is an N-methyl-D-aspartic acid receptor antagonist with potent analgesic and sedative properties. Evidence suggested that esketamine could be used as a component of sedative regimen in many settings, such as endoscopy and endoscopic retrograde cholangiopancreatography. Nevertheless, there remains an evidence gap in the efficacy and safety of esketamine used in bronchoscopy. Therefore, we conducted this study to test the hypothesis that low-dose esketamine as an adjuvant to propofol was non-inferior to propofol alone on the recovery profile and discharge from the hospital after ambulatory bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) classification I-III;
2. Scheduled for ambulatory bronchoscopy.

Exclusion Criteria:

1. Allergic or contraindications to studying drugs
2. History of obstructive sleep apnea-hypopnea syndrome
3. History of psychiatric illness
4. History of neurological disease
5. Pre-existing memory or cognitive impairment
6. History of seizure disorders
7. Pregnancy
8. Substance abuse or intake of drugs that affect the central nervous system
9. Inability to communicate in Mandarin Chinese.
10. Illiteracy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Proportions of patients discharged within 30 min after bronchoscopy | Up to 40 minutes postoperatively
  Discharge readiness will be measured using the Modified Post Anesthetic Discharge Scoring System scale (greater than or equal to nine).

SECONDARY OUTCOMES:
Postoperative quality of recovery | Baseline, up to 72 hours postoperatively
  Postoperative quality of recovery will be measured using the Postoperative Quality of Recovery Scale (PostopQRS). The PostopQRS is a digital measurement tool to quantify physiological, emotive, nociceptive, activities of daily living, and cognitive domain of postoperative recovery over time. Recovery in various domains of the PostopQRS is defined by postoperative values equaling or exceeding individual baseline values.
Injection pain | Immediately after administering the study drugs, on average 2 minutes
  Injection pain was assessed using a numeric rating scale of 0 to 10 (0 equals no pain, and 10 equals the worst pain imaginable).
Emergency time | Immediately after the bronchoscopy completely withdrawn, on average 8 minutes
  Emergency time was defined as the interval from the end of bronchoscopy to the MOAA/S score equal to five.
Incidence of adverse events | Up to 72 h postoperatively
  Episodes of adverse events such as bradycardia, tachycardia, hypotension, hypertension, hypoxia, nausea, vomiting, nightmare, and blurred vision
Propofol consumption | During the bronchoscopy procedure
  Propofol consumption will be recorded during the bronchoscopy procedure.
Patient willingness to repeat the procedure | 24 hours postoperatively
  Patients will be asked whether they would repeat the identical procedural process (Yes/No/Unsure).
Bronchoscopist satisfaction | At completion of bronchoscopy procedure
  Bronchoscopist satisfaction will be evaluated using a five-point Likert scale (5=very satisfied, 4=satisfied, 3=neither satisfied nor dissatisfied, 2=dissatisfied, and 1=very dissatisfied).
Patient satisfaction | At completion of bronchoscopy procedure
  Bronchoscopist satisfaction will be evaluated using a five-point Likert scale (5=very satisfied, 4=satisfied, 3=neither satisfied nor dissatisfied, 2=dissatisfied, and 1=very dissatisfied).
Patient willingness to recommend screening | 24 hours postoperatively
  Patients will be asked whether they would recommend bronchoscopy screening to a friend or a relative (Yes/No/Unsure).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaochun Zheng, MD, Study Chair — Fujian Provincial Hospital
Locations (1):
- Fujian provincial hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
After publication, the individual deidentified participant data underlying published results, the study protocol, and the statistical analysis plan can be accessed upon reasonable request from the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: We would like to share our individual deidentified participant data beginning three months following the publication of the main results.
Access Criteria: All of the individual participant data collected during the trial, the study protocol, the statistical analysis plan, and the clinical study report can be accessed with approval from the corresponding author.